CLINICAL TRIAL: NCT02768363
Title: A Randomized Controlled Trial Of AdV-tk + Valacyclovir Administered During Active Surveillance For Newly Diagnosed Prostate Cancer
Brief Title: Randomized Controlled Trial of CAN-2409 Immunotherapy During Active Surveillance for Prostate Cancer (ULYSSES)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Candel Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PrTK04
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: Immunotherapy; Tumor vaccine; Immuno-oncology; Cytotoxicity; Prostate cancer; Active Surveillance
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAN-2409 (Active Comparator): Patients randomized to the active arm will receive two courses of aglatimagene besadenovec (CAN-2409) + valacyclovir
  Interventions: Biological: aglatimagene besadenovec; Drug: valacyclovir
- Placebo (Placebo Comparator): Patients randomized to the placebo arm will receive two corresponding courses of placebo + valacyclovir
  Interventions: Biological: placebo; Drug: valacyclovir

INTERVENTIONS:
Biological: aglatimagene besadenovec — Aglatimagene besadenovec will be delivered to the prostate via trans-rectal ultrasound guided injection followed by 14 days of oral prodrug, valacyclovir. The second aglatimagene besadenovec injection will be 2-3 weeks after the first followed by 14 days of valacyclovir.
  Other Names: AdV-tk; CAN-2409
  Arms: CAN-2409
Biological: placebo — Placebo will be delivered to the prostate via trans-rectal ultrasound guided injection followed by 14 days of oral prodrug, valacyclovir. The second placebo injection will be 2-3 weeks after the first followed by 14 days of valacyclovir.
  Arms: Placebo
Drug: valacyclovir — Oral prodrug to be given for 14 days starting the day after each aglatimagene besadenovec or placebo injection.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of CAN-2409 immunotherapy in patients undergoing active surveillance for localized prostate cancer. CAN-2409 involves the use of aglatimagene besadenovec to kill tumor cells and stimulate a cancer vaccine effect. Killing tumor cells in an immune stimulatory environment induces the body's immune system to detect and destroy cancer cells. CAN-2409 has been well tolerated in previous trials in patients with prostate cancer and other tumor types. Biochemical, pathologic and immune responses have been demonstrated in newly diagnosed and recurrent prostate cancer. The hypothesis is that CAN-2409 can lead to improvement in the clinical outcome for patients with prostate cancer. Participants will be randomized to the CAN-2409 or control arm at a 2:1 ratio. Both arms receive standard of care active surveillance evaluations.

ELIGIBILITY:
Inclusion Criteria include:

* Histologically confirmed adenocarcinoma of the prostate
* Patients choosing active surveillance
* Patients meeting definition of NCCN low risk, intermediate risk OR patients having only one NCCN high-risk feature

  * NCCN Low Risk is defined as having all of the following: PSA < 10 ng/ml, Gleason ≤ 6, T1-T2a
  * NCCN Intermediate Risk is defined as having at least one of the following and no high risk features: PSA 10-20 ng/ml, Gleason score =7, T2b-T2c
  * High Risk with a single high risk feature is defined as having only one of the following: PSA>20 ng/ml, Gleason score 8-10, or T3a
  * Excluded are those in the following risk groups: High risk with more than 1 high risk factor; Locally advanced/very high risk=T3b-T4; Metastatic: N1 or M1
* Patients must be planning and medically able to tolerate multiple transrectal ultrasound guided injections.
* ECOG Performance status 0-2

Exclusion Criteria include:

* Active liver disease, including known cirrhosis or active hepatitis
* Patients on systemic corticosteroids (>10 mg prednisone per day) or other immunosuppressive drugs
* Known HIV+ patients
* Regional lymph node involvement or distant metastases
* Other current malignancy (except squamous or basal cell skin cancers)
* Other serious co-morbid illness or compromised organ function that, in the opinion of the investigator, would interfere with treatment or follow up
* Prior treatment for prostate cancer except TURP. If prior TURP, patients must be deemed able to receive prostate biopsy and multiple intra-prostatic injections by the investigator
* Patients taking 5-alpha-reductase inhibitors (e.g. finasteride, dutasteride)
* Patients who had or plan to use ADT or have history of an orchiectomy.
* Patients who are planning to undergo radical treatment for prostate cancer within 12 months.
* Known sensitivity or allergic reactions to acyclovir or valacyclovir

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2016-05; Primary Completion 2024-11 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Baseline to study completion, approximately 5 years
  Progression-free survival is defined as the time from randomization to evidence of histological disease progression or death due to prostate cancer

SECONDARY OUTCOMES:
Negative biopsy rate at 1-year landmark | 1 year
Percentage of patients with adverse events | 30 days after last dose of study drug

CONTACTS AND LOCATIONS:
Locations (23):
- United States (22):
  - Foothills Urology, Golden, Colorado
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Southeast Louisiana Veterans Health Care System, New Orleans, Louisiana
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Sierra Nevada Health Care System VA, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Advanced Radiation Centers of New York (Integrated Medical Professionals), North Hills, New York
  - Associated Medical Professionals of NY, PLLC, Syracuse, New York
  - Southwest Urology, Clinical Research Solutions, Middleburg Heights, Ohio
  - Oklahoma City VA Healthcare System, Oklahoma City, Oklahoma
  - VA Portland Health Care System, Portland, Oregon
  - Oregon Urology Insitute, Springfield, Oregon
  - Lancaster Urology, Lancaster, Pennsylvania
  - Allegheny Health Network-Triangle Urological Group, Pittsburgh, Pennsylvania
  - Ralph H. Johnson Veterans Affairs Medical Center, Charleston, South Carolina
  - San Antonio VA Healthcare System, San Antonio, Texas
  - Woodland Center, The Woodlands, Texas
  - Texas Urology Specialists, Tomball, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Salem VA Medical Center, Salem, Virginia
- Instituto Nacional de Ciencias Medicas y Nutrición, Salvador Subirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No